CLINICAL TRIAL: NCT06223308
Title: A Phase I/II Open Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of HB0028 in Patients With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety and Efficacy of HB0028 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0028-01
Record Dates: First submitted 2023-12-24; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A single-subject cohort will be enrolled at the protocol starting dose of HB0028 every 3 weeks (Q3W). Dose escalation will proceed to the next main dose level according to the 3+3 dose-escalation procedure until the MTD/OBD is reached. Phase II of the study will be initiated at the Sponsor's discretion at the dose level and treatment schedule which was established as the recommended Phase 2 dose (RP2D) in the dose-escalation phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HB0028 (Experimental): HB0028 IV every 3 weeks (q3w)
  Interventions: Drug: HB0028

INTERVENTIONS:
Drug: HB0028 — Patients will be assigned to dose regimens in the order of enrollment, and they will receive their assigned fixed dose of HB0028 via intravenous infusion. HB0028 IV every 3 weeks (q3w).
  Other Names: Anti-PD-L1 and TGF-β bifunctional fusion protein

SUMMARY:
It is a phase I/II open label, multicenter study to assess the safety, tolerability, pharmacokinetics, and efficacy of HB0028 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase I/II, multicenter, open-label, first-in-human study in patients with advanced solid tumors. During the phase I study, the safety and tolerability of HB0028 will be evaluated in patients with advanced solid tumors. In the phase II study, the safety and efficacy of HB0028 at the RP2D will be evaluated in cohorts of patients with specific solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria to be eligible for participation in this study:

  1. Male or female. Age ≥ 18 years.
  2. The subject is able to understand and willing to sign the Informed Consent Form(ICF); willing and able to comply with all study procedures.
  3. a) dose escalation: Patients with histologically or cytologically confirmed locally advanced, recurrent, or metastatic solid tumors (or clinically diagnosed hepatocellular carcinoma) that failed all standard therapies known to provide clinical benefit; [These solid tumors include but not limit to: non-small cell lung cancer, esophageal squamous cell carcinoma, melanoma, head and neck squamous cell carcinomas, hepatocellular carcinoma, gastric or gastroesophageal junction adenocarcinoma, renal cell carcinoma, etc.].

     b) dose expansion (Cervical cancer group): Histologically confirmed persistent, recurrent, or metastatic ([International Federation of Gynecology and Obstetrics(FIGO)] stage IVB) cervical cancer that is not eligible for curative surgery and/or definitive concurrent radiotherapy; The pathological type was squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma.; According to the investigator's judgment, it may benefit from the study drug treatment; patients with disease progression after at least one previous systemic therapy (such as systemic chemotherapy).
  4. At least one measurable tumor lesion was present according to RECIST 1.1. A baseline imaging assessment could be performed up to 28 days before the first dose.
  5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
  6. Life expectancy ≥12 weeks
  7. liver function requirements:

     1. Total bilirubin (TBIL) ≤ 1.5×ULN
     2. Aspartate aminotransferase(AST) and Alanine aminotransferase(ALT) ≤ 2.5×ULN; AST or ALT ≤5×ULN if liver metastases are present;
  8. Creatinine (Scr) < 1.5×ULN and Calculated creatinine clearance (CrCL) > 50 mL/ min (Cockroft-Gault Equation);
  9. Hematology absolute neutrophil count (ANC) ≥ 1.5×109/L; hemoglobin (HGB) ≥ 90 g/L ；platelets (PLT) ≥ 75×109/L;
  10. Coagulation function: International Normalized Ratio(INR)≤ 1.5×ULN; Prothrombin Time(PT)≤ 1.5×ULN; Activated Partial Thromboplastin Time(APTT)≤ 1.5×ULN. No active or clinically significant bleeding within 14 days before the first dose.
  11. Recovery to Grade 0-1 from adverse events (AEs) related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, and endocrinopathies controlled with hormone replacement therapy
  12. Women of childbearing potential must confirm a negative serum or urine pregnancy test within 3 days prior to the initiation of study treatment; Fertile patients and their partners must agree to use effective contraceptives for the duration of study drug use and for 90 days after the last administration of study treatment.

Exclusion Criteria:

* Exclusion Criteria Patients are excluded from the study if any of the following criteria apply:

  1. Have clinically active central nervous system (CNS) metastases. Patients with previously-treated brain or meningeal metastases may participate and be eligible for treatment provided they are stable (>4 weeks) and asymptomatic. Patients with asymptomatic brain metastasis or subjects who are symptomatically stable after treatment and are on < 10 mg/d prednisone or equivalent are eligible.
  2. dose expansion (Cervical cancer group): Hydronephrosis, which could not be relieved by clinical treatment
  3. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
  4. History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for grade 3 endocrinopathy that is managed with hormone replacement therapy).
  5. Use of systemic corticosteroids in a dose equivalent to >10 mg/day of prednisone or other immunosuppressive agent < 2 weeks prior to screening; the use of topical, intraocular, intraarticular, intranasal, or inhaled corticosteroids and systemic steroids to prevent (e.g., allergy to contrast agents) or treat non-autoimmune condition (e.g., delayed hypersensitivity caused by exposure to allergens) or short course (< 5 days) will be allowed
  6. Cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure < 6 months of study entry; uncontrolled arrhythmia < 3 months of study entry; mean ECG QT-interval corrected according to Fridericia's formula (QTcF) > 470 milliseconds (ms) obtained from three ECGs;
  7. uncontrolled diabetes, glycosylated hemoglobin HbA1c >8%；
  8. Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (According to RECIST v1.1).
  9. Patients who have previously received allogeneic stem cell, Bone marrow or solid organ transplantation.
  10. The following infections are present

      1. Active infection requiring intravenous treatment within 2 weeks before screening
      2. Active Pulmonary tuberculosis
      3. Positive results for HIV test
      4. Active hepatitis B or C. Patients with asymptomatic hepatitis B virus carriers (HBV DNA titer < 1000 cps/mL or 200 IU/mL) or cured hepatitis C virus(HCV)(negative HCV RNA test) may be enrolled;
  11. Major surgery < 4 weeks prior to the first dose; Minor surgery < 2 weeks prior to the first dose
  12. History of severe allergic reactions, grade 3-4 allergic reactions to treatment with another monoclonal antibody, or known to be allergic to protein drugs or recombinant proteins or excipients in HB0028 drug formulation;
  13. Have received or will receive a live vaccine within 30 days prior to the screening.
  14. Patients who have participated in any clinical trial of a drug or medical device within 30 days prior to the first dose
  15. Any other serious underlying medical condition (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), or psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment.
  16. Positive COVID-19 quantitative real time (qRT) polymerase chain reaction (PCR) or rapid screening test during screening;
  17. Patients with a history of arterial or deep vein thrombosis within 6 months before enrollment; evidence or history of a bleeding tendency within 2 months before enrollment
  18. Severe dyspnea, pulmonary insufficiency or the need for continuous supportive oxygen therapy
  19. The surgical site, the wound site, the mucous membrane severely ulcerated, or the fracture did not heal completely
  20. Conditions that may cause bleeding or perforation of the digestive tract (such as duodenal ulcer, intestinal obstruction, Crohn's disease, Ulcerative colitis, large gastrectomy and small bowel resection, etc.); Patients with a history of intestinal perforation and fistula, who were not cured after surgical treatment; Esophageal and gastric varices
  21. Immunomodulatory therapy was administered within 2 weeks before enrollment (including but not limited to cyclosporine and tacrolimus)
  22. Have history of interstitial lung disease or non-infectious pneumonitis, except from radiotherapy (the enrollment of subjects needs to be considered after discussion with MM);
  23. Other conditions which would make it inappropriate for the patient to participate as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 12 Months
  Number of participants with a Dose Limiting Toxicity(DLT)[Time Frame:During the first days]DLTs will be assessed during the first 21 days of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria,and assessed as having a suspected or definite relationship to study drug.
Maximun Tolerated Dose(MTD) | Up to 24 Months
  MTD or Optimal Biological Dose(OBD) and/or RP2D.

SECONDARY OUTCOMES:
AUC | Up to 24 Months
  AUC Area Under concentration-time Curve (AUC)
Cmax | Up to 24 Months
  Maximum serum concentration(Cmax)
Tmax | Up to 24 Months
  Half-life time of maximum concentration
ORR | Up to 24 Months
  Overall response rate(ORR) as measured by RECIST v1.1.

OTHER OUTCOMES:
Percentage of the lymphocyte subpopulations. | Up to 24 Months
  The percentage of lymphocyte subpopulations of the peripheral blood will be assessed by flow cytometry.
Programmed death ligand 1(PDL1) expression level | Up to 24 Months
  The expression of PD-L1 in tumor tissues was detected by immunohistochemical method.
Tubuloglomerular Feedback(TGF-β) | Up to 24 Months
  Levels of TGF-β1, TGF-β2, TGF-β3 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD/PHD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No